CLINICAL TRIAL: NCT01807013
Title: Prospective Study to Evaluate the Diagnostic Value of B-mode Ultrasound, Elastometry and Minilaparoscopic Guided Liver Biopsy for the Diagnosis of Compensated Liver Cirrhosis.
Brief Title: Evaluating Ultrasound, Elastometry, Minilaparoscopy and Histology for the Diagnosis of Compensated Liver Cirrhosis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital Erlangen (Other)
Responsible Party: Principal Investigator, Prof. Dr. D. Strobel, Prof. Dr., University Hospital Erlangen
Other Study IDs: LapSon
Record Dates: First submitted 2012-07-12; First posted 2013-03-08 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Cirrhosis
Keywords: cirrhosis; liver; elastometry; ultrasound; laparoscopy; diagnosis
MeSH Terms: conditions — Fibrosis; Disease | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: ultrasound, liver elastometry, minilaparoscopy — * conventional high-end ultrasound technique,
  * small access laparoscopy with fine laparoscopes
  * Acoustic radiation force impulse (ARFI): ARFI technology uses short-duration acoustic radiation forces (approximately 100 microseconds) to generate a localized tissue displacement which results in a lateral shear-wave propagation. ARFI shear wave velocity (SWV) measured in m/sec tracked with ultrasonic correlation-based methods is proportional to the square root of tissue elasticity.

SUMMARY:
Prospective study to evaluate the dignostic value of b-mode ultrasound, elastometry and mini-laparoscopic guided liver biopsy for the diagnosis of compensated liver cirrhosis.

DETAILED DESCRIPTION:
Up to now the gold standard for the diagnosis of liver cirrhosis is to perform liver biopsy. This invasive methode is not undisputed. Therefore there is constant effort to improve, develop and apply better diagnostic tools. This study is designed to evaluate the in our eyes now a days most promising examinations: (1) high frequency ultrasound, (2) elastometry and (3) minilaparoscopy. Patients for whom the clinical decision to perform mini laparoscopic guided liver biopsy was taken should be recruited. Successive at three time points the examiner has to decide for or against cirrhosis: (1) after conventional and high frequency ultrasound (2) after elastometry and (3) after laparoscopy.

ELIGIBILITY:
Inclusion Criteria:

* clinical decision to perform minilaparoscopic guided liver biopsy for the staging of liver disease including the assessment of the degree of fibrosis.

Exclusion Criteria:

* ascites
* decompensated liver disease
* esophageal varices
* other collateral circulations
* obstructive cholestasis
* severe heart insufficiency (NYHA III-IV)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with suspected chronic liver disease
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-02; Primary Completion 2014-08 (Actual); Study Completion 2016-08 (Estimated)

PRIMARY OUTCOMES:
Prospective Evaluation of Acoustic Radiation Force Impulse (ARFI) Elastography and High-Frequency B-Mode Ultrasound in Compensated Patients for the Diagnosis of Liver Fibrosis/Cirrhosis in Comparison to Mini-Laparoscopic Biopsy | blood tests, b-mode ultrasound, ARFI and minilaparoscopy to be done preferential within 48 hours
  Histology is obtained at minilaparoscopy. For an Ishak fibrosis stage of 5/6 or a clearly nodular liver surface at minilaparoscopy cirrhosis is confirmed.

SECONDARY OUTCOMES:
Can the non invasive tests be combined resulting in a better accuracy for the prediction of liver cirrhosis/fibrosis? | blood tests, b-mode ultrasound, ARFI and minilaparoscopy to be done preferential within 48 hours

OTHER OUTCOMES:
What liver related complications develop and by which test are they best predicted? | Follow up patients for 3/5 years

CONTACTS AND LOCATIONS:
Overall Officials: Deike Stobel, Prof. Dr., Study Director — Universitätsklinikum Erlangen-Nürnberg
Locations (1):
- Universitätsklinikum Erlangen Nürnberg, Erlangen, Bavaria, Germany